CLINICAL TRIAL: NCT04108026
Title: A Phase II Single-arm Trial Evaluating Safety and Efficacy of Durvalumab in ECOG Performance Status 2-3, Treatment-naive, Patients With Stage IV Non-Small Cell Lung Cancer (NSCLC) and High PD-L1 Tumor Expression
Brief Title: Immunotherapy in Patient With Poor General Condition
Acronym: SAVIMMUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1802
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer Stage IV
Keywords: IFCT; Savimmune; Non small cell Lung Cancer; PS; Poor General condition; Lung Cancer; Durvalumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immunotherapy (Experimental): Durvalumab 1500 mg every 4 weeks until the progression of disease, discontinuation due to toxicity or withdrawal of consent, for a maximum duration of 2 years.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — 1500 mg IV every 4 weeks

SUMMARY:
Immunotherapeutic approaches targeting immune checkpoint proteins PD-1/PD-L1 have recently demonstrated clinical efficacy in several cancer types, and have changed the therapeutic landscape in metastatic melanoma or non-small cell lung cancer (NSCLC).

The monoclonal anti-PD-1 antibody nivolumab has been registered by both FDA (Food and Drug Administration) and EMA (European Medicine Agency), for metastatic NSCLC patients, after failure of a prior platinum-based chemotherapy.

The approval was based on the results of phase III clinical trials in metastatic NSCLC. But all the trials only enrolled patients with good general condition, PS (Performance Status) 0 or 1. However, the prevalence of poor PS patients at time of diagnosis is high in lung cancer patients.

For patients with metastatic NSCLC and PS 3, there is no standard treatment except best supportive care, since all trials that accrued unselected PS 3 patients fail to prove any survival advantage, and most PS >3 patients die within 2 to 4 months from diagnosis. Indeed, these patients are currently excluded from clinical trials. Specific dedicated clinical trials and treatment guidelines for this patient population are urgently needed, taking into account for the high prevalence of such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an IEC (Independent Ethic Committee) approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.

   Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
2. Histologically or cytologically-proven NSCLC (squamous or non-squamous). If the diagnosis is cytologically-proven, sufficient material is necessary with at least 100 tumor cells evaluated for PD-L1 IHC (Immunohistochemistry).
3. PD-L1 expression ≥25% of tumor cells as assessed by the local pathology laboratory using protocols validated.
4. Available tumor samples for centralized PD-L1 immunohistochemistry analysis.
5. No EGFR (Epidermal Growth Factor Receptor) mutation and no ALK(Anaplasic Lymphoma Kinase) gene rearrangement.
6. Stage IV (8th classification TNM) M1a or M1b or M1c.
7. ECOG (Eastern Cooperative Oncology Group) PS = 2 or 3 despite optimal symptomatic treatment.
8. Body weight >30kg
9. No prior systemic anticancer therapy (chemotherapy, immunotherapy including durvalumab, or EGFR or ALK inhibitors) given as primary therapy for advanced or metastatic disease. Neoadjuvant or adjuvant chemotherapy is not considered as chemotherapy for advanced or metastatic disease.
10. Limited field of radiation for palliation within 2 weeks of the first dose of durvalumab is allowed, provided the lung is not in the radiation field and irradiated lesion(s) cannot be used as target lesions.
11. Age 18-75 years.
12. Measurable tumor disease by CT per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
13. Life expectancy > 8 weeks according to the investigator opinion.
14. Adequate biological functions:

    neutrophils ≥ 1500/mm3 ; platelets ≥ 75 000/mm3 ; Hemoglobin ≥ 9 g/dL ; Creatinine Clearance > 40 mL/min , AST and ALT ≤ 2,5 ULN unless liver metastases are present, AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤ 5 x ULN, serum bilirubin ≤ 1.5 x ULN except for patients with proved, Gilbert syndrome (≤ 5 x ULN) or patients with hepatic metastases (≤ 3 x ULN).
15. Other investigations detailed in Section 5 must have been performed within the timelines indicated.
16. Protocol treatment is to begin within 7 days of patient inclusion.
17. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
18. Females of childbearing potential who are sexually active with a nonsterilized male partner or men who are sexually active with women of childbearing potential must use a highly effective method of contraception prior the first dose of investigational product, and must agree to continue using such precautions for 90 days after the final dose of investigational product. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

1. Pure or combined SCLC.
2. Known HER2 (Human Epidermal Growth Factor Receptor), B-Raf, activating tumor mutations, or exon 14 c-MET splice mutations (mesenchymal-epithelial transition), or known ROS1 gene rearrangement.
3. Asymptomatic or symptomatic brain metastasis.
4. Carcinomatous meningitis.
5. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with IFCT
   * Patients with celiac disease controlled by diet alone
6. Immunosuppressive treatment including systemic treatment with corticosteroids with greater dose than 10 mg prednisone equivalent daily, within 15 days before enrollment. Inhaled, nasal or topic corticosteroids are allowed.
7. History of allogenic organ transplantation.
8. Stage 4 (very severe, FEV1 (forced expiratory volume at one second) <30% predicted) chronic obstructive pulmonary disease (COPD) according to GOLD classification.
9. NYHA (New York Heart Association) class 4 chronic heart failure
10. Pre-existing interstitial lung.
11. History of another primary malignancy except for :

    * Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IP (Investigational Product) and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of residual disease Patients with a prostate adenocarcinoma history within the previous 5 years could be included in case of localized prostate cancer.
12. Living attenuated vaccine received within the 30 previous days.
13. Received any other experimental treatment or participation to any other therapeutic clinical trial.
14. Known allergy or hypersensitivity to any of the study drug or any of the study drug excipients.
15. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
16. Major surgical procedure within 28 days prior to the first dose of IP or planned surgical procedure during treatment.
17. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs (Adverse Events) or compromise the ability of the patient to give written informed consent.
18. Active infection including tuberculosis, hepatitis B (known positive HBV surface antigen (HBsAg) result) and hepatitis C,. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. History of active tuberculosis or evident primo-infection for which there is no record or evidence of an active anti-tuberculous treatment (please consult IFCT in case of doubt).
19. Patient with human immunodeficiency virus (positive HIV ½ antibodies)
20. Any condition that, in the opinion of investigator, could compromise the adherence to treatment and follow-up.
21. Mental illness or psychological condition, which in the opinion of investigator could compromise the expression of the informed consent.
22. No public health insurance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing Grade 3-5 Treatment Related Adverse Event at 8 weeks of durvalumab | 8 weeks

SECONDARY OUTCOMES:
Incidence, type and severity of adverse event | From time of informed consent through treatment period (24 months) or up to 100 days post last dose of study treatment
  The maximum grade will be summarized by frequency and proportion of total patients, by system organ class and NCI-CTC, Version 5.0 categories.
Disease Control Rate | 8 weeks
  Percentage of patients with objective response or stable disease according to RECIST 1.1 in the intent to treat population
Objective Response Rate according to BICR (Blinded Independent Central Review) and investigators | 8 weeks (confirmed at 16 weeks)
  Percentage of patients with objective response according to RECIST 1.1 in the intent to treat population
Progression free survival | 6 and 12 months
  Time between the date of durvalumab initiation and the first date of documented progression or death due to any cause, whichever occurs first.
Overall survival | 6 and 12 months
  Time between the date of durvalumab initiation and the date of death due to any cause, whichever occurs first.
Performance status improvement rate | From time of randomisation through treatment period (24 months)
  Proportion of per-protocol patients whose PS during durvalumab treatment was improved from baseline
Evaluate the Quality of life | From time of randomisation through treatment period (24 months)
  EORTC QLQ-C30 +LC13 (Qualify of Life Questionnaire C30 + Lung Cancer 13) questionnaire
Centrally-assessed PD-L1 tumor expression Prognostic and predictive value | Baseline only
Evaluate the Quality of life | From time of randomisation through treatment period (24 months)
  EQ-5D (EuroQol 5 Dimensions) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Valérie GOUNANT, Study Chair — AP-HP Hôpital Bichat-Claude Bernard; Michael DURUISSEAUX, Study Chair — Hospices Civils de Lyon - Hôpital Louis Pradel
Locations (20):
- France (20):
  - Besançon - CHU, Besançon
  - Hôpital Ambroise Paré - Pneumologie, Boulogne
  - Caen - CHU Côte de Nacre, Caen
  - CH, Colmar
  - CHRU Grenoble, Grenoble
  - Centre Hospitalier - Pneumologie, Le Mans
  - CHRU de Lille, Lille
  - AP-HM Hopital Nord, Marseille
  - Montpellier - CHRU, Montpellier
  - GRH Mulhouse Sud-Alsace, Mulhouse
  - Nancy - Institut de Cancérologie de Lorraine, Nancy
  - Nantes - ICO Site René Gauducheau, Nantes
  - CHR d'Orléans La Source, Orléans
  - AP-HP Hopital Tenon - Pneumologie, Paris
  - Paris - APHP Bichat, Paris
  - Paris - Curie, Paris
  - Lyon - URCOT, Pierre-Bénite
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse - Pneumologie, Toulouse
  - CHU Tours - Pneumologie, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: IFCT website — http://www.ifct.fr